CLINICAL TRIAL: NCT06729905
Title: Study of the Effects of Yerba Mate on Cardiometabolic Health
Acronym: INFU-SALUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Ciencia y Tecnología de Alimentos y Nutrición (Other Government)
Collaborators: Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AGL2010-18269
Record Dates: First submitted 2024-12-07; First posted 2024-12-12 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Risk; Hypercholerolemia
Keywords: Yerba mate; Cardiovascular health; Inflammation; Blood lipids; Glucose homeostasis
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yerba mate (Experimental): Consumption of three cups of a yerba mate tea per day
  Interventions: Dietary Supplement: Yerba mate tea
- Control (Other): Consuming water or an isotonic drink, free of polyphenols or caffeine.
  Interventions: Dietary Supplement: Control drink

INTERVENTIONS:
Dietary Supplement: Yerba mate tea — Consumption of three cups per day of a beverage prepared with yerba mate
  Arms: Yerba mate
Dietary Supplement: Control drink — Consumption of water or an isotonic drink, free of polyphenols or caffeine. Abstention of consuming coffee.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if consuming a beverage prepared with yerba mate leaves helps to improve blood lipid levels in persons at high cardiovascular risk. It will also learn about the effects of this beverage, widely consumed in South America, on other cardiometabolic biomarkers like blood glucose levels, inflammation, or weight control. The main questions it aims to answer are:

Does daily consumption of a yerba mate tea reduce the blood lipid levels in hypercholesterolemic persons? May healthy persons also benefit from the consumption of yerba mate tea?

Researchers will compare yerba mate to a control drink (isotonic drink or water, free of polyphenols and caffeine) to see if yerba mate tea helps to reduce blood cholesterol in hypercholesterolemic persons.

Participants will:

Drink 3 cups of yerba mate tea or an isotonic drink every day for 2 months, then change to the other drink during another 2 months.

Visit the clinic at the beginning and end of each 2-month period for checkups and tests Refraing from consuming coffee and some foods during the study. Complete a dietary questionnaire during 3 days before each visit to the clinic.

DETAILED DESCRIPTION:
This is a randomized, crossover, control study in healthy and hypercholesterolemic free-living to assess the effect of yerba mate on different outcomes related to cardiovascular health.

After a 2-week run-in period, participants will be randomly allocated to the first 8-weeks intervention with yerba mate or the control drink. After a 3-week wash-out, they will change to consume during 8 weeks the other drink.

A nurse will collect a fasting blood sample at the beginning and end of each intervention stage. Blood pressure and anthropometric parameters will be measured. A 72-h dietary record will be completed by participants before each visit to the Human Nutrition Unit (HNU) at the Institute of Food Science, Technology and Nutrition (ICTAN-CSIC).

During the study, participants will refrain from consuming coffee, cocoa, tea, and caffeine-containing drinks. Other foods rich in certain polyphenols (i.e. hydroxycinnamic acids) will also be restricted.

Blood samples will be used to measure different biomarkers of relevance in cardiometabolic health, as listed in the Outcomes section.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 20-25 kg/m2
* Total cholesterol < 200 mg/dL for healthy participants, between 200-240 mg/dL for participants at cardiovascular risk, or
* LDL cholesterol < 130 mg/dL for healthy participants, between 130-159 mg/dL for participants at cardiovascular risk.

Exclusion Criteria:

* Smoking
* Pregnant/lactating women
* Vegetarians/vegans
* Consumption of vitamins or dietary supplements
* Suffering from chronic diseases/pathologies/conditions appart from hypercholesterolemia
* On prescription drugs (statins) or on antibiotics 6 months before the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-01-10 (Actual); Primary Completion 2013-07-30 (Actual); Study Completion 2015-05-30 (Actual)

PRIMARY OUTCOMES:
Blood lipids | From enrollment to the end of each treatment at 8 weeks
  Change in blood levels of total cholesterol or LDL-cholesterol or VLDL-cholesterol or HDL-cholesterol or triglycerides or phospholipids at the end of the intervention with yerba mate

SECONDARY OUTCOMES:
Blood pressure | From enrollment to the end of each treatment at 8 weeks
  Changes in blood pressure at the end of the intervention with yerba mate.
Inflammatory cytokines | From enrollment to the end of each treatment at 8 weeks
  Change in the levels of C-reactive protein (CRP), or pro-inflammatory cytokines (tumor necrosis factor-alpha (TNF-a), or interferon gamma (IFN-g), interleukin (IL)-1beta (IL-1b), or IL-2, or IL-5, or IL-6, or IL-7, or IL-8, or IL-12 or IL-13)) or anti-inflammatory cytokines IL-4 or IL-10 at the end of the intervention with yerba mate
Fasting blood glucose | From enrollment to the end of each treatment at 8 weeks
  Change of fasting blood glucose levels at the end of the intervention with yerba mate
Fasting blood insulin | From enrollment to the end of each treatment at 8 weeks
  Change of fasting insulin levels at the end of intervention with yerba mate
Insulin resistance | From enrollment to the end of each treatment at 8 weeks
  Change in homeostasis model assessment (HOMA) of insulin resistance (HOMA-IR) at the end of intervention with yerba mate
Insulin sensitivity | From enrollment to the end of each treatment at 8 weeks
  Change in quantitative insulin levels sensitivity check index (QUICKI) at the end of the intervention with yerba mate. Higher score in QUICKI means a better outcome compared to initial values.
Hormones, incretins and adipokines levels | From enrollment to the end of each treatment at 8 weeks
  Changes in serum levels of C peptide or glucagon or glucagon inhibitory peptide (GIP) or glucagon-like peptide type 1 (GLP-1) or ghrelin or leptin or resistin or plasminogen activator inhibitor type 1 (PAI-1) or visfatin at the end of the intervention with yerba mate.
Cytokines, chemokines and cell-adherence molecules levels | From enrollment to the end of each treatment at 8 weeks
  Changes in serum levels of granulocyte (G-CSF) or granulocyte/macrophague (GM-CSF) colony-stimulating factors, or monocyte-chemoattractant protein-1 (MCP-1) or macrophage inflammatory protein-1beta (MIP-1b) or vascular (VCAM-1) or intracellular (ICAM-1) adhesion molecules at the end of the intervention with yerba mate.
Liver function | From enrollment to the end of each treatment at 8 weeks
  No changes in serum levels of alanin transferase (ALAT), or aspartate transferase (ASAT) at the end of the intervention with yerba mate.
Anthropometry | From enrollment to the end of each treatment at 8 weeks
  Changes in body weight or body fat percentage or body circunferences (wais, or hip, or thigh, or brachial) or skinfolds (tricipital or subscapular) at the end of the intervention with yerba mate.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bravo, Professor, Principal Investigator — ICTAN-CSIC
Locations (1):
- Instituto de Ciencia y Tecnología de Alimentos y Nutrición, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bravo L, Martinez-Lopez S, Sierra-Cinos JL, Mateos R, Sarria B. Yerba Mate (Ilex paraguariensis St. Hill.) Tea May Have Cardiometabolic Beneficial Effects in Healthy and At-Risk Subjects: A Randomized, Controlled, Blind, Crossover Trial in Nonhabitual Consumers. Mol Nutr Food Res. 2025 Aug;69(15):e70065. doi: 10.1002/mnfr.70065. Epub 2025 Apr 22. PMID 40263915